CLINICAL TRIAL: NCT00236613
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group, Dose-Response Study to Assess the Efficacy and Safety of Topiramate in the Treatment of Patients With Obesity
Brief Title: A Study on Efficacy and Safety of Topiramate in the Treatment of Patients With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003709
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Obesity
Keywords: Obesity; Hypertension; Hyperlipidemia; Body Mass Index
MeSH Terms: conditions — Obesity; Hypertension; Hyperlipidemias | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of topiramate (64mg, 96mg, 192mg, and 384mg daily) with placebo in the treatment of obesity.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. This is a randomized, double-blind, placebo-controlled, multicenter study to assess the safety and effectiveness of topiramate in treatment of obese patients. Patients will receive 24 weeks of treatment by topiramate or placebo, followed by 2 week taper and a safety follow-up. Effectiveness will be determined by changes from baseline to week 24 in body weight, body mass index (BMI), anthropometric measurements (waist circumference, hip circumference, waist/hip ration), fasting lipid profiles, fasting plasma glucose, HbA1c (shows average blood sugar level over months), fasting uric acid, fasting insulin, and blood pressures. Safety evaluations (incidence of adverse events, physical examinations, 12 lead ECGs, vital signs, Computerized Neuropsychological Test Battery) will be performed throughout the study. The study hypothesis is that topiramate will be effective in achieving and maintaining weight reduction in obese patients and is well tolerated. The patients will be randomized to receive either topiramate (64, 96, 192, or 384 mg daily) or placebo daily by mouth for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >=30 and <50
* BMI >= 27 and < 50 if patient has controlled hypertension or abnormal blood lipids
* Stable weight
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Known contraindication, or hypersensitivity to topiramate
* Exposure to any other experimental drug or device within last 30 days
* A diagnosis of diabetes
* History or evidence of clinically significant liver disease, cardiovascular disease, uncontrolled hypertension or high thyroid levels
* History of obesity with known cause
* History or family history of kidney stones
* History of weight loss surgery
* History of malignancy within last 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2000-09; Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
The percent change in body weight from baseline (at the time of randomization) to Week 24.

SECONDARY OUTCOMES:
Changes from baseline to week 24 in total body weight, body mass index, fasting plasma glucose; incidence of adverse events over study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Bray GA, Hollander P, Klein S, Kushner R, Levy B, Fitchet M, Perry BH. A 6-month randomized, placebo-controlled, dose-ranging trial of topiramate for weight loss in obesity. Obes Res. 2003 Jun;11(6):722-33. doi: 10.1038/oby.2003.102. PMID 12805393
- [Derived] Loring DW, Williamson DJ, Meador KJ, Wiegand F, Hulihan J. Topiramate dose effects on cognition: a randomized double-blind study. Neurology. 2011 Jan 11;76(2):131-7. doi: 10.1212/WNL.0b013e318206ca02. Epub 2010 Dec 9. PMID 21148119